CLINICAL TRIAL: NCT07118995
Title: Anatomical Feasibility of the Braile Off-the-Shelf Multi-Branched Endograft for the Treatment of Thoracoabdominal Aneurysm
Brief Title: ANATOMICAL FEASIBILITY OF BRAILE STANDARD BRANCHED ENDOGRAFT
Acronym: BMETA
Status: Active, not recruiting | Type: Observational
Sponsor: Braile Biomedica Ind. Com. e Repr. Ltda. (Industry)
Responsible Party: Sponsor
Other Study IDs: BMETA
Record Dates: First submitted 2025-08-05; First posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Thoracoabdominal Aortic Aneurysm; Endovascular Repair of Aortic Aneurysm; Vascular Diseases; Aortic Diseases; Aortic Aneurysm
Keywords: Thoracoabdominal aortic aneurysm; Off-the-shelf endograft; Anatomical feasibility
MeSH Terms: conditions — Aortic Aneurysm, Thoracoabdominal; Vascular Diseases; Aortic Diseases; Aortic Aneurysm

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients treated for TAA: Patients with thoracoabdominal aortic aneurysms treated with a custom-designed multi-branched endograft.
  Interventions: Other: Analysis of preoperative CTA

INTERVENTIONS:
Other: Analysis of preoperative CTA — A review of preoperative contrast-enhanced CTA from patients with thoracoabdominal aneurysms, included in Braile's database, who were indicated for endovascular treatment with Braile's custom-made multi-branched endograft between 2022 and 2024

SUMMARY:
The objective of this retrospective observational study is to evaluate the theoretical anatomical suitability of the new Braile off-the-shelf multi-branched endograft in patients with thoracoabdominal aneurysm. One hundred preoperative contrast-enhanced computed tomography angiographies (CTAs) from patients previously treated with a custom-made endograft will be analyzed. The hypothesis is that a significant proportion of these patients will have anatomical features compatible with the use of the new endograft.

ELIGIBILITY:
Inclusion Criteria:

* Preoperative CTA images from patients previously treated with Braile's custom-made multi-branched endograft for thoracoabdominal aneurysm.
* Contrast-enhanced CTAs covering the thorax, abdomen, and pelvis, with thin slices of 1 to 2 mm, available in Braile's imaging database.

Exclusion Criteria:

• Exams with incomplete or inadequate images, defined as CTAs with slice thickness greater than 2 mm

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with thoracoabdominal aortic aneurysm
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2025-08-01 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Anatomical feasibility and applicability of off-the-shelf multi-branched endografts from two device models | completion of the anatomical assessment
  Number of patients with anatomical characteristics suitable for the theoretical use of the new Braile off-the-shelf multi-branched endograft.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre A Pereira, Principal Investigator — Hospital Moinho de Ventos
Locations (1):
- Hospital Moinho de Ventos, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No